CLINICAL TRIAL: NCT00674921
Title: Cotrimoxazole Prophylaxis Cessation Study Among Stabilized HIV-Infected Adult Patients on HAART in Entebbe, Uganda
Acronym: CCS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Dr George Miiro, MRC/UVRI Uganda Research Unit on Aids
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 009/ESR/NDA/DID-01/2008
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: Opportunistic Infections; AIDS; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): It will comprise patients randomized to receive the placebo (stop cotrimoxazole prophylaxis) at CD4 counts of 200 or more but less than 350 cells/ul as they continue with HAART. Patients will be followed until they achieve a CD4 count of 350 cells/ul.
  Interventions: Drug: Placebo
- 2 (Active Comparator): It will comprise patients randomized to continue with cotrimoxazole prophylaxis and HAART at CD4 counts of 200 or more but less than 350 cells/ul. These patients will be followed until they achieve a CD4 count of 350 cells/ul and above, at which point they will be considered for the second randomization.
  Interventions: Drug: cotrimoxazole
- A (Placebo Comparator): This arm will comprise patients who have achieved a CD4 count of 350 or more cells/ul either at the beginning of the study or once they have reached this threshold at the end of follow up in arms 1 and 2. They (including those previously in Arm 1) will receive the placebo (stop cotrimoxazole prophylaxis) after the second randomization but continue with HAART.
  Interventions: Drug: Placebo
- B (Active Comparator): It will comprise patients randomized to continue or start with cotrimoxazole prophylaxis and HAART at CD4 of 350 or more cells/ul after second randomization. Some of them will have used cotrimoxazole prophylaxis whilst they were in arm 2 and others in arm 1 will restart cotrimoxazole prophylaxis at this stage.
  Interventions: Drug: cotrimoxazole

INTERVENTIONS:
Drug: cotrimoxazole — cotrimoxazole 800/160 mg once daily as indicated by the start and end times of the specified arms for continued prevention of HIV-related infections
  Arms: 2; B
Drug: Placebo — starch, magnesium stearate, sodium lauryl sulphate
  Arms: 1; A

SUMMARY:
According to the national guidelines in Uganda and to the World Health Organization guidelines, HIV-infected patients should receive cotrimoxazole prophylaxis indefinitely. There are, however, concerns regarding the indefinite application of cotrimoxazole prophylaxis among patients immunologically stabilized on HAART (e.g. high pill burden, drug-drug interactions, toxicity and poor adherence because of treatment fatigue). To date no empirical evidence is available regarding the safety and optimal timing for the cessation of cotrimoxazole prophylaxis among HAART patients who successfully restored immunological competence.

Research question: Does morbidity significantly differ between continuation (orthodox) and cessation (experimental) of cotrimoxazole prophylaxis among immuno-competent patients stable HAART in the resource-limited setting of Uganda?

DETAILED DESCRIPTION:
Randomized double-blind placebo controlled equivalence trial to be conducted among consenting clinically healthy patients on HAART with 2 or more CD4 counts of 200 cells/ul or more for at least 3 months. The study will enable comparison of effects of randomized cessation of cotrimoxazole prophylaxis at 2 CD4-guided thresholds (200 Vs 350 cells/ul).

Rationale for inclusion of the placebo-controlled design

* The double-blind placebo controlled approach is feasible and ethically justified in this equipoise situation to allow for concealment of allocated intervention among investigators and patients and avoids accidental unblinding of investigators to the allocated interventions by trial patients.
* Maintenance of continued cotrimoxazole prophylaxis among patients randomized to this intervention will be easier if there is no awareness that those patients randomized to cessation of prophylaxis have a relative advantage of reduced pill burden.
* It would be very difficult to maintain cessation of cotrimoxazole prophylaxis among patients randomized to do so in our setting where cotrimoxazole is readily and cheaply available in drug shops, drug stores and pharmacies.

First randomisation

Patients who have been on HAART for at least 3 months and who have a confirmed CD4 count between 200 and 349 cells/ul will be randomized to continue prophylaxis with active cotrimoxazole or to cease prophylaxis with active cotrimoxazole but continue with ingestion of the placebo cotrimoxazole daily.

Second randomization

Patients who achieve a confirmed CD4 count of 350 cells/ul or more while on HAART will be randomized to continue prophylaxis with active cotrimoxazole or to cease prophylaxis with active cotrimoxazole but continue with ingestion of placebo cotrimoxazole daily. Some patients will have participated already in 1st randomization but others will be entering the trial at this stage for the first time.

Rationale for 4 trial arms

In order to assess the separate effects of cessation of cotrimoxazole prophylaxis in trial patients at the 2 randomization stages above, those continuing with prophylaxis will be compared with those ceasing prophylaxis, necessitating 2 arms at each stage.

ELIGIBILITY:
Inclusion Criteria:

* Consenting HIV-infected patient aged 16 years or older,
* Resident within 40 kms of study clinics
* Regularly attending clinics
* Documented HAART intake for at least 3 months
* Clinically healthy and stable
* Confirmed CD4 count of 200 cells/ul more.

Exclusion Criteria:

* Acutely ill patients with opportunistic or other infections
* Patients already enrolled in other HAART trials (e.g DART trial)
* First trimester pregnancy at enrolment
* Clinical and immunological evidence of HAART treatment failure
* Unable to attend study clinics regularly
* Hypersensitivity to cotrimoxazole

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1650 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
all-cause morbidity such as pneumonia or malaria (presumptive and definitive diagnosis) | 3 years

SECONDARY OUTCOMES:
sub-clinical laboratory abnormalities (such as neutropenia) and serious adverse events (such as death) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: George Miiro, MSc, MBChB, Principal Investigator — MRC/UVRI Unit; Heiner Grosskurth, PhD, MD, Study Director — MRC/UVRI Unit; Paula Munderi, MRCP, MBChB, Principal Investigator — MRC/UVRI Unit
Locations (1):
- MRC/UVRI Uganda Research Unit on Aids, Entebbe, Uganda

REFERENCES:
- [Result] Zellweger C, Opravil M, Bernasconi E, Cavassini M, Bucher HC, Schiffer V, Wagels T, Flepp M, Rickenbach M, Furrer H; Swiss HIV Cohort Study. Long-term safety of discontinuation of secondary prophylaxis against Pneumocystis pneumonia: prospective multicentre study. AIDS. 2004 Oct 21;18(15):2047-53. doi: 10.1097/00002030-200410210-00009. PMID 15577626
- [Result] Mussini C, Pezzotti P, Antinori A, Borghi V, Monforte Ad, Govoni A, De Luca A, Ammassari A, Mongiardo N, Cerri MC, Bedini A, Beltrami C, Ursitti MA, Bini T, Cossarizza A, Esposito R; Changes in Opportunistic Prophylaxis (CIOP) Study Group. Discontinuation of secondary prophylaxis for Pneumocystis carinii pneumonia in human immunodeficiency virus-infected patients: a randomized trial by the CIOP Study Group. Clin Infect Dis. 2003 Mar 1;36(5):645-51. doi: 10.1086/367659. Epub 2003 Feb 12. PMID 12594647
- [Result] Ledergerber B, Mocroft A, Reiss P, Furrer H, Kirk O, Bickel M, Uberti-Foppa C, Pradier C, D'Arminio Monforte A, Schneider MM, Lundgren JD; Eight European Study Groups. Discontinuation of secondary prophylaxis against Pneumocystis carinii pneumonia in patients with HIV infection who have a response to antiretroviral therapy. Eight European Study Groups. N Engl J Med. 2001 Jan 18;344(3):168-74. doi: 10.1056/NEJM200101183440302. PMID 11188837
- [Result] Esposito S, Bojanin J, Porta A, Cesati L, Gualtieri L, Principi N. Discontinuation of secondary prophylaxis for Pneumocystis pneumonia in human immunodeficiency virus-infected children treated with highly active antiretroviral therapy. Pediatr Infect Dis J. 2005 Dec;24(12):1117-20. doi: 10.1097/01.inf.0000190038.53813.d2. PMID 16371882
- [Result] Lopez Bernaldo de Quiros JC, Miro JM, Pena JM, Podzamczer D, Alberdi JC, Martinez E, Cosin J, Claramonte X, Gonzalez J, Domingo P, Casado JL, Ribera E; Grupo de Estudio del SIDA 04/98. A randomized trial of the discontinuation of primary and secondary prophylaxis against Pneumocystis carinii pneumonia after highly active antiretroviral therapy in patients with HIV infection. Grupo de Estudio del SIDA 04/98. N Engl J Med. 2001 Jan 18;344(3):159-67. doi: 10.1056/NEJM200101183440301. PMID 11172138
- [Result] Furrer H, Egger M, Opravil M, Bernasconi E, Hirschel B, Battegay M, Telenti A, Vernazza PL, Rickenbach M, Flepp M, Malinverni R. Discontinuation of primary prophylaxis against Pneumocystis carinii pneumonia in HIV-1-infected adults treated with combination antiretroviral therapy. Swiss HIV Cohort Study. N Engl J Med. 1999 Apr 29;340(17):1301-6. doi: 10.1056/NEJM199904293401701. PMID 10219064
- [Result] Weverling GJ, Mocroft A, Ledergerber B, Kirk O, Gonzales-Lahoz J, d'Arminio Monforte A, Proenca R, Phillips AN, Lundgren JD, Reiss P. Discontinuation of Pneumocystis carinii pneumonia prophylaxis after start of highly active antiretroviral therapy in HIV-1 infection. EuroSIDA Study Group. Lancet. 1999 Apr 17;353(9161):1293-8. doi: 10.1016/s0140-6736(99)03287-0. PMID 10218526